CLINICAL TRIAL: NCT03917069
Title: Nab-paclitaxel Plus Carboplatin Combined Endostatin Versus Solvent-based Paclitaxel Plus Carboplatin in the Treatment of Advanced Melanoma After the Failure of PD-1 Treatment #A Randomized Controlled, Open, Multicenter Trial
Brief Title: Nab-PCE vs PC for MM After Failure of Anti-PD-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun GUO, Vice President of Beijing Cancer Hospital，Head of renal carcinoma & melanoma dept., Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019NPCE
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Advanced Melanoma
Keywords: nab-paclitaxel; carboplatin; endostatin; melanoma
MeSH Terms: conditions — Melanoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nab-paclitaxel + endostatin+ carboplatin (Experimental): nab-paclitaxel + endostatin+ carboplatin nab-paclitaxel 260mg/m2, d1 +Carboplatin AUC=5, d1 +endostatin 15mg, d1-14 q28d
  Interventions: Drug: Chemotherapeutic Combinations
- paclitaxel+carboplatin (Active Comparator): paclitaxel+carboplatin paclitaxel 175 mg/m2, d1+ Carboplatin AUC=5, d1 q21d
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: Chemotherapeutic Combinations — nab-paclitaxel 260mg/m2 d1+Carboplatin AUC=5 d1+ endostatin 15mg d1-14，q28d
  Arms: nab-paclitaxel + endostatin+ carboplatin
Drug: chemotherapy — paclitaxel 175 mg/m2 d1+Carboplatin AUC=5 d1, q21d
  Arms: paclitaxel+carboplatin

SUMMARY:
This is a randomized controlled clinical trial of nab-paclitaxel + carboplatin

* Endostatin for advanced melanoma after failure of PD-1 therapy. The aim was to evaluate the efficacy and safety of nab-paclitaxel+carboplatin
* endostatin versus combination of paclitaxel and carboplatin in patients with advanced melanoma after failure of PD-1 therapy.

DETAILED DESCRIPTION:
The enrollment time is expected to be 1.5 year and the observation time is 2 years. The regimen were performed on a 28-day/21-day cycle respectively. Subjects who met the entry criteria were treated in a 2:1 group according to a randomized list: the treatment group was treated with nab-paclitaxel + carboplatin + endostatin regimen, and the control group was treated with paclitaxel + carboplatin. In this trial, the efficacy is evaluated every 8 weeks until disease progression or unacceptable toxicity,or until the investigator deemed that the patient's condition was unacceptable for further treatment. The follow-up period was 24 months after the end of treatment (follow-up patient survival information and new anti-tumor treatment). The planning enrolled sample size for nab-paclitaxel + carboplatin + endostatin group and paclitaxel-carboplatin group were 90 patients and 45 patients, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 70 years old, male or female;
2. Histological or pathological diagnosis of advanced melanoma, and progressed after anti-PD-1 treatment (disease progression or unacceptable toxicity);
3. The patient has at least one (RECIST 1.1 standard) measurable lesion, which needs to be detected by spiral CT or MRI, and the tumor lesion has at least one single diameter ≥ 1 cm;
4. ECOG PS is 0 or 1 (see Annex 1 for standards);
5. The estimated survival period is ≥12 weeks;
6. no chemotherapy contraindications, including normal peripheral blood, liver and kidney function and electrocardiogram are basically normal; Peripheral blood: neutrophils ≥1.5×109/L, platelets≥90×109/ L, hemoglobin≥90 g/L; Renal function: normal serum creatinine; For patients with non-metastatic liver function impairment: alanine, aspartate aminotransferase ≤ 2.5 ULN, For patients with metastatic liver dysfunction: alanine, aspartate aminotransferase ≤ 5 ULN;
7. Patients who have undergone topical treatment for asymptomatic brain metastases can be enrolled and have a clinical stable status of at least 4 weeks.
8. Patients voluntarily participate in and sign an informed consent form.
9. contraindications for the use of no carboplatin, paclitaxel, entropic and albumin paclitaxel

Exclusion Criteria:

1. Known HIV, hepatitis B/C virus positive status or history of active tuberculosis (testing prior to randomisation is not required)
2. Received any investigational drug within 28 days or 5 half-lives of the planned first dose of this study treatment.
3. Active infection requiring systemic therapy.
4. A known history of another malignancy or concurrent malignancy unless the patient is disease-free for a minimum of 1 year, is completely treated and is at low-risk of recurrence.
5. Patients with a history or evidence of cardiovascular risk,
6. History or evidence of interstitial lung disease or active non-infectious pneumonitis.
7. Serious or unstable pre-existing medical conditions or other conditions that could interfere with the patient's safety, consent, or compliance.
8. Pregnant or breastfeeding females, or expecting to conceive or father children within the projected period of study treatment (52 weeks followed by 4 months following end of study treatment).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2019-03-23 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 3 years
  The time from treatment to tumor progression or death

SECONDARY OUTCOMES:
Objective response rate (ORR) | At the end of Cycle 2 (each cycle is 28 days)
  response evaluation disease progression defined by Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) criteria.
  response (PR), refers to the number of cases with complete and partial response after treatment as a percentage of the total number of evaluable cases
Disease Control Rate (DCR) | At the end of Cycle 2 (each cycle is 28 days)
  The disease control rate was the proportion of patients with complete remission, partial remission and stability (SD) in all patients.
overall survival (OS) | 3 years
  OS was defined as the time from the date of the first administration of trial regimen to the date of death from any cause (event) or last follow-up (censored data).
Adverse events (AE) | 3 years
  Adverse events (AE) were monitored on an ongoing basis and classified according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0. Patients were assessed for toxicities before each administration, and toxicity was graded accordingly

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Dr., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: data access requests will be reviewed by an external Independent Review Panel.Requestors will be required to sign a Data Access Agreement.
URL: http://www.guojun.org/